CLINICAL TRIAL: NCT03360227
Title: Registry of Device Implantation in University Hospital Duesseldorf
Brief Title: Registry of Device Implantation
Status: Recruiting | Type: Observational
Sponsor: Klinik für Kardiologie, Pneumologie und Angiologie (Other)
Responsible Party: Sponsor-Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Principal Investigator, Heinrich-Heine University, Duesseldorf
Organization: Heinrich-Heine University, Duesseldorf (Other)
Other Study IDs: 15-019
Record Dates: First submitted 2017-11-08; First posted 2017-12-04 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Syncope; Bradycardia; Tachycardia; Sudden Cardiac Death; Ventricular Tachycardia; Ventricular Fibrillation
Keywords: syncope; bradycardia; tachycardia; sudden cardiac death; implantable cardioverter-defibrillator; ventricular tachycardia; ventricular fibrillation; biomarker; thyroid hormone
MeSH Terms: conditions — Syncope; Bradycardia; Tachycardia; Death, Sudden, Cardiac; Tachycardia, Ventricular; Ventricular Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

INTERVENTIONS:
Device: implantation of cardiac devices — implantation of cardiac devices

SUMMARY:
The implantable device therapy for cardiac arrhythmias has been an established therapy, and one of the common standard procedures in cardiac clinical practice.

Pacemakers, implantable cardioverter-defibrillators, and cardiac resynchronization therapy have been developed since 1960s, and the technologies in this field are still progressively developing. Not only these "traditional" implantable devices, there are multiple new devices for cardiac diseases, such as implantable loop recorder, vagal nerve stimulator and barostimulator.

The aim of this registry is to demonstrate the efficacy and the safety of standard device implantation procedures and to evaluate/ identify specific factors, including clinical characteristics, laboratory data and procedural data, which predict the prognosis/complication of the patients. These identification will result in further improvement of patients' care.

DETAILED DESCRIPTION:
The implantation of cardiac devices has been one of the common standard procedures in the cardiac clinical practice.

Pacemakers are implanted for patients with symptomatic bradyarrhythmias. Implantable cardioverter-defibrillators are implanted in order to avoid sudden cardiac death (SCD) in high risk patients such as after myocardial infarction and reduced ejection fraction.

Cardiac resynchronization therapy was introduced to improve the prognosis in patients with reduced EF and left bundle branch block. This therapy demonstrated the efficacy in severe heart failure patients.

Recently a new implantable device has been developed also to improve the prognosis of patients with severe heart failure refractory to the maximal therapies at present. This barostimulator activates the baro-reflex and results in higher parasympathetic activity and better outcome in those patients, in whom the sympathetic function is overactivated.

In patients with cryptogenic stroke or syncope, the implantable loop recorder enables us to monitor the cardiac rhythm continuously for 3 years. With this device, the occult arrhythmias can be revealed and lead patients to the adequate therapy.

Above mentioned device therapies have been developed since 1960s, and the technologies in this field are still progressively developing. To catch up these advancements, the quality management including the efficacy, safety aspects and the prognosis of the patients should be carefully monitored.

The aim of the present study is, therefore, to demonstrate the efficacy and the safety of standard device implantation procedures. The patient specific and procedural factors are evaluated to test if those factors predict the prognosis of the patients. These identifications will eventually result in the improvement of future patients' care.

The data of patients who underwent device implantation since 2011 and those who undergo device implantation till 2019 will be collected, including the basic demographic data, comorbidities, results of laboratory and functional tests. In the latter patients, the peri-procedural data and post-procedural data are also prospectively collected.

The present study is essentially an observational study. The inclusion in this study does not affect the decision of device implantation itself. The post-procedural therapies, such as medications and device therapies are not due to this registry affected.

As a sub-project in this registry, biomarkers and thyroid hormone are evaluated to investigate the predictable value of those indices.

ELIGIBILITY:
Inclusion Criteria:

1. pre-operative clinical history taking
2. pre-operative functional investigations (cardiac echo, electrocardiograms)
3. pre-operative laboratory data evaluation (kidney function, liver function, biomarkers, thyroid hormone, CBC)

Exclusion Criteria:

１. no written informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergo cardiac device implantation in University Hospital Düsseldorf
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2011-01 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
device related adverse events | during index hospital admission
  Adverse events as occurrence of perioperative and postoperative complication related to the device implantation during the index hospital admission
Adverse Events | during index hospital admission
  Adverse Events as occurrence of atrial fibrillation, occurrence of syncope, occurrence of sustained ventricular tachycardia (VT), ventricular fibrillation (VF) or appropriate ICD therapy including antitachycardia pacing (ATP) and shock, occurrence of inadequate ICD therapy including ATP and shock in ICD/CRT-D patients, hospital admission due to cardiac disease and therapy, cardiac death

SECONDARY OUTCOMES:
survival | 12 months
Clinical Events | 12 months
  free from clinical events (death, syncope, hospital admission due to cardiac problems, and VT storm [defined as more than three VT episodes in 24 hours])
hospitalization | 12 months
  hospitalization due to cardiac disease and therapy
number of appropriate and inappropriate ICD therapies (ATP or shock) | 12 months
  number of appropriate and inappropriate ICD therapies (ATP or shock)

CONTACTS AND LOCATIONS:
Overall Officials: Hisaki Makimoto, MD, Principal Investigator — Division of Cardiology, Pulmonary Disease and Vascular Medicine
Locations (1):
- Division of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf, Germany